CLINICAL TRIAL: NCT03865550
Title: Evaluation of Post Operative Pain Following Primary Total Knee Arthroplasty (TKA) With Intraoperative Subanesthetic Ketamine Administration and Spinal Anesthesia
Brief Title: Post-op Ketamine Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Rothman Institute Orthopaedics (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016Levicoff
Record Dates: First submitted 2019-03-05; First posted 2019-03-07 (Actual); Last update posted 2019-03-07 (Actual); Status verified 2019-03

CONDITIONS: Osteo Arthritis Knee
MeSH Terms: interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Isotonic saline
- Ketamine (Active Comparator)
  Interventions: Drug: Ketamine Injectable Solution

INTERVENTIONS:
Drug: Isotonic saline — Placebo
  Arms: Placebo
Drug: Ketamine Injectable Solution — Active comparator
  Arms: Ketamine

SUMMARY:
The purpose of this study is to establish the effect of sub-anesthetic dosing of ketamine with spinal anesthesia during total knee arthroplasty on post-operative pain and narcotic consumption. We hypothesize that sub-anesthetic ketamine will decrease post-operative pain and narcotic consumption and may secondarily lead to shorter lengths of stay, faster rehabilitation, improved postoperative outcomes and patient satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 years of age
* ASA I - IV
* Undergoing primary unilateral elective total knee arthroplasty with spinal anesthesia

Exclusion Criteria:

* BMI over 40*
* Contraindication or allergy to opioid pain medication or ketamine*
* Daily opioid use for pain control before surgery in excess of systemic morphine equivalent to 10 mg*
* Ejection fraction (EF) less than 30%
* Creatinine clearance less than 30 mL/min*
* History of chronic liver failure
* Desire for nerve block or general anesthesia
* Any neurologic or psychiatric disorder (including bipolar disorder, post traumatic stress disorder, schizophrenia)
* Prior surgery on ipsilateral knee within the last 6 months
* Alcohol abuse

Age Groups: Child, Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2016-03-28 (Actual); Primary Completion 2018-04-27 (Actual); Study Completion 2019-04-27 (Estimated)

PRIMARY OUTCOMES:
Pain as reported on Visual Analog Scale | Up to 6 weeks post-operatively
  VAS pain reported 0-100mm

CONTACTS AND LOCATIONS:
Locations (1):
- Rothman Institute, Philadelphia, Pennsylvania, United States